CLINICAL TRIAL: NCT07367152
Title: Predictors of Treatment Success After Intercostal Nerve Radiofrequency for Intercostal Neuralgia: A Retrospective Cohort Study
Brief Title: Predictors of Success After Intercostal Nerve Radiofrequency Treatment for Intercostal Neuralgia
Acronym: ICN-RF-IN
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mesut Bakır, Associate Professor, Mersin University
Other Study IDs: MERSINALG-INTERCOSTALRF-2026
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Intercostal Neuralgia; Postherpetic Neuralgia ( PHN ); Thoracic Neuropathic Pain
Keywords: Intercostal nerve; Pulsed radiofrequency; Conventional radiofrequency; Ultrasound-guided
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intercostal Nerve Radiofrequency Cohort: Adults with intercostal neuralgia who underwent ultrasound-guided intercostal nerve radiofrequency treatment (conventional or pulsed) as part of routine clinical care.
  Interventions: Procedure: Intercostal Nerve Conventional Radiofrequency Ablation (CRF); Procedure: Intercostal Nerve Pulsed Radiofrequency (PRF)

INTERVENTIONS:
Procedure: Intercostal Nerve Conventional Radiofrequency Ablation (CRF) — Ultrasound-guided intercostal nerve lesioning at 80°C for 90 seconds following sensory stimulation.
Procedure: Intercostal Nerve Pulsed Radiofrequency (PRF) — Ultrasound-guided intercostal pulsed radiofrequency delivered at 42°C for 240 seconds.

SUMMARY:
This retrospective cohort study will review medical records of patients treated with intercostal nerve radiofrequency for intercostal neuralgia. The goal is to identify patient and clinical factors that are associated with treatment success after the procedure. Outcomes will be assessed using pain measures documented during routine follow-up visits, along with any recorded adverse events. No additional visits, tests, or interventions are required because this study uses previously collected clinical data.

DETAILED DESCRIPTION:
This retrospective cohort study analyzed anonymized medical records of adults (≥18 years) with intercostal neuralgia (post-traumatic, postherpetic, or idiopathic) treated in Pain Clinic of Mersin University Faculty of Medicine who underwent ultrasound-guided intercostal conventional radiofrequency ablation (CRF) or pulsed radiofrequency (PRF) between January 1, 2018 and May 30, 2025.

Primary outcome is treatment response at 6 months, defined by IMMPACT criteria as a ≥50% reduction or ≥4-point decrease in NRS-11 from baseline; secondary outcomes include changes in NRS-11 over time, and exploratory analyses evaluate whether clinical factors (e.g., age, sex, pain duration, diagnosis, presence of allodynia, and number of treated intercostal levels )are associated with response using multivariable logistic regression (p < 0.05 considered statistically significant).

The findings are expected to clarify which patient and clinical characteristics are linked to better outcomes after intercostal nerve radiofrequency and to support more individualized decision-making in the management of intercostal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of intercostal neuralgia (post-traumatic, postherpetic, or idiopathic) with thoracic neuropathic pain for at least 1 month
* Underwent ultrasound-guided intercostal nerve radiofrequency treatment (conventional radiofrequency ablation [CRF] or pulsed radiofrequency [PRF]) as part of routine clinical care
* Documented baseline NRS-11 pain score prior to the procedure and follow-up NRS-11 data available through at least 6 months after treatment.

Exclusion Criteria:

* Thoracic pain attributable to malignancy-related causes (e.g., active malignant invasion, spinal metastasis) or an intrathoracic mass
* History of thoracic surgery at the corresponding thoracic dermatome level (e.g., thoracotomy or VATS)
* Prior radiofrequency treatment at the same intercostal nerve site
* Receipt of other interventional treatments targeting the intercostal nerve during the study period (e.g., cryoablation or chemical neurolysis)
* Insufficient follow-up data (less than 6 months of follow-up NRS-11 documentation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with intercostal neuralgia who underwent ultrasound-guided intercostal nerve radiofrequency treatment (conventional or pulsed) in routine clinical care and had documented baseline and at least 6-month follow-up NRS-11 pain scores.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Treatment response at 6 months (IMMPACT-defined responder rate) | 6 months
  Responder defined as ≥50% reduction or ≥4-point decrease in NRS-11 compared with baseline.

SECONDARY OUTCOMES:
Change in NRS-11 pain score from baseline | Baseline, 3 months, and 6 months
  NRS-11 ranges from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Medicine, Department of Algology, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective study based on de-identified patient records. No individual participant data (IPD) will be shared. Only aggregated results may be published in scientific journals.

REFERENCES:
- [Result] Huang X, Ma Y, Wang W, Guo Y, Xu B, Ma K. Efficacy and safety of pulsed radiofrequency modulation of thoracic dorsal root ganglion or intercostal nerve on postherpetic neuralgia in aged patients: a retrospective study. BMC Neurol. 2021 Jun 24;21(1):233. doi: 10.1186/s12883-021-02286-6. PMID 34162352
- [Result] Engel AJ. Utility of intercostal nerve conventional thermal radiofrequency ablations in the injured worker after blunt trauma. Pain Physician. 2012 Sep-Oct;15(5):E711-8. PMID 22996865